CLINICAL TRIAL: NCT07166458
Title: Fuctional Assessment of Kefir Fermented Milk on the Improvement of Osteoporosis Combined With Fracture Patient
Brief Title: Kefir Peptides for Bone Fracture Healing
Acronym: KPs-Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jen-Chieh Lai (Other)
Responsible Party: Sponsor-Investigator, Jen-Chieh Lai, Taichung Armed Forces General Hospital, National Chung Hsing University
Organization: National Chung Hsing University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B202005023
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Bone Fractures
MeSH Terms: conditions — Fractures, Bone | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two parallel groups: one group receiving kefir peptide supplementation plus standard care, and the other group receiving standard care alone.
Who Masked: Participant, Care Provider
Masking Description: Participants and care providers are blinded to treatment assignment. The kefir peptide supplement and placebo are identical in appearance and packaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kefir Peptide + Standard Care (Experimental): Participants will receive kefir peptide supplementation in addition to standard fracture care.
  Interventions: Dietary Supplement: Kefir Peptide
- Standard Care (Active Comparator): Participants will receive standard fracture care without kefir peptide supplementation.
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Dietary Supplement: Kefir Peptide — Oral supplementation with kefir-derived bioactive peptides given daily in addition to standard care.
  Arms: Kefir Peptide + Standard Care
Other: Standard Care (in control arm) — Standard fracture management including immobilization, pain control, and routine follow-up care.
  Arms: Standard Care

SUMMARY:
This study is designed to evaluate the effects of kefir-derived peptides on bone healing in patients with upper limb fractures. Kefir peptides are natural protein fragments that may promote bone formation and reduce inflammation. Participants with recent upper limb fractures will be randomly assigned to receive either kefir peptide supplementation or standard treatment. The main purpose of this study is to determine whether kefir peptides can accelerate bone healing and improve recovery compared to standard care.

DETAILED DESCRIPTION:
This study aims to investigate the efficacy of kefir-derived peptides in enhancing bone healing after upper limb fractures. Kefir peptides are bioactive fragments of milk proteins that have shown potential in stimulating osteoblast differentiation, inhibiting osteoclast activity, and modulating inflammation in preclinical studies.

The study is designed as a randomized, controlled clinical trial. Eligible participants with acute upper limb fractures will be randomly assigned to receive either kefir peptide supplementation in addition to standard care, or standard care alone. The primary objective is to evaluate radiographic and clinical healing at 6 months, while secondary outcomes include pain relief, functional recovery, and quality of life measures.

This trial seeks to provide clinical evidence supporting kefir peptides as a safe and natural adjunct therapy to accelerate bone repair, potentially reducing recovery time and improving functional outcomes for patients with fractures.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients with a bone mineral density T-score determined by dual energy X-ray absorptiometry (DXA) < -2.5 or patients with acute fragile fractures in the distal radius and proximal humerus, and additionally (2) women with menopause or (3) patients who are over 50 years of age.

Exclusion Criteria:

* (1) a body mass index (BMI) > 30, (2) those who have been administered pharmacological agents such as glucocorticoids, thyroxine, antiepileptics, bisphosphonates, calcitonin, and hormone replacement therapy, or medications impacting bone metabolism for a duration over 4 months, and (3) individuals with a documented medical history of hyperparathyroidism, hyperthyroidism, diabetes mellitus, hepatic cirrhosis, and renal insufficiency

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Radiographic Healing Score at 3 Months | 3 months after fracture fixation
  Bone healing will be assessed using standard radiographs and the modified Lane and Sandhu scoring system.

CONTACTS AND LOCATIONS:
Locations (1):
- National Chung Hsing University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lai JC, Chang GR, Tu MY, Cidem A, Chen IC, Chen CM. Potential of Kefir-Derived Peptides, Probiotics, and Exopolysaccharides for Osteoporosis Management. Curr Osteoporos Rep. 2025 Apr 7;23(1):18. doi: 10.1007/s11914-025-00910-9. PMID 40192921
- [Background] Lai JC, Li HP, Chang GR, Lan YW, Chen YH, Tseng YS, Tu MY, Chen CF, Chen HL, Chen CM. Kefir peptides promote osteogenic differentiation to enhance bone fracture healing in rats. Life Sci. 2022 Dec 1;310:121090. doi: 10.1016/j.lfs.2022.121090. Epub 2022 Oct 17. PMID 36257457
- See also: Related Info — https://www.nchu.edu.tw